CLINICAL TRIAL: NCT07403487
Title: A Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial to Evaluate the Efficacy and Safety of RC1416 Injection in Adult Patients With Moderate to Severe Asthma
Brief Title: Phase II Trial of RC1416 Injection in Asthma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing RegeneCore Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RJK-RC1416-103
Record Dates: First submitted 2026-01-27; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Moderate to Severe Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RC1416 (Experimental)
  Interventions: Drug: RC1416
- RC1416 Placebo (Placebo Comparator)
  Interventions: Drug: RC1416 Placebo

INTERVENTIONS:
Drug: RC1416 — There are two doses in this part. Each subjects will receive the drug by subcutaneous injection.
  Arms: RC1416
Drug: RC1416 Placebo — Each subjects will receive the placebo by subcutaneous injection
  Arms: RC1416 Placebo

SUMMARY:
This study is a phase II study of RC1416 in subjects with severe uncontrolled asthma. The purpose of the study is to evaluate efficacy and safety of RC1416 in subjects with severe uncontrolled asthma.

DETAILED DESCRIPTION:
RC1416 is a bispecific homodimer nanobody .It is being developed by Nanjing RegeneCore Biotech Co., Ltd. as a potential therapy for asthma. A total 195 severe uncontrolled asthma subjects will be enrolled in three groups to access the efficacy and safety of RC1416.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and 75 years.
* Diagnosed with asthma for at least 1 year, and the current disease status meets the diagnostic criteria of the 2024 GINA guidelines.
* Have received medium-to-high dose ICS therapy for at least 3 consecutive months prior to screening, and maintained a stable treatment regimen and dose for ≥1 month prior to baseline.
* Pre-bronchodilator forced expiratory volume in 1 second (FEV1) measurement ≤80% of the predicted normal value at both the screening and baseline visits.
* Asthma Control Questionnaire-6 (ACQ-6) score ≥1.5 at both the screening and baseline visits.
* Must have experienced ≥1 severe asthma exacerbation event within the 12 months prior to screening.
* Positive bronchodilator reversibility test.

Exclusion Criteria:

* Individuals with a known history of allergy to the investigational product or its excipients.
* Clinically diagnosed with chronic obstructive pulmonary disease (COPD) or other lung diseases that may impair lung function .
* Experienced a severe asthma exacerbation event from within 1 month prior to screening until before dosing.
* Used systemic corticosteroids within 1 month prior to screening.
* Had a pulmonary or other site infection requiring intravenous antibiotics, antifungals, or antivirals from within 1 month prior to screening until before dosing.
* Used traditional Chinese medicine with anti-asthmatic effects within 1 month prior to screening.
* Underwent major surgery within 8 weeks prior to screening or plans to undergo major surgery during the study period.
* With a history of malignancy within the past 5 years .
* Active or incompletely treated tuberculosis
* Used biologic/systemic immunosuppressant/immunomodulators within 12 weeks or 5 half-lives prior to screening.
* Diagnosed active parasitic infection; suspected parasitic infection or high risk of infection.
* Abnormal 12-lead electrocardiogram (ECG) at screening. The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Estimated)
Dates: Start 2026-03-10 (Estimated); Primary Completion 2027-10-25 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Pre-bronchodilator (Pre-BD) forced expiratory volume in 1 Second (FEV1) | During 32 weeks
  Mean change from baseline in Pre-BD forced expiratory volume in 1 Second (FEV1)

SECONDARY OUTCOMES:
Severe asthma exacerbation | During 32 weeks
  Severe asthma exacerbation events, Time to the first asthma exacerbation
Pre-BD FEV1 | During 32 weeks
Morning and evening peak expiratory flow (PEF) | During 32 weeks
  Mean change from baseline of absolute value and percentage
forced vital capacity (FVC) | During 32 weeks
  Mean change from baseline of absolute value and percentage
Forced mid-expiratory flow (FEF25-75%) before bronchodilator (BD) | During 32 weeks
  Mean change from baseline of absolute value and percentage
Asthma loss of control (LOAC) | During 32 weeks
  Asthma loss of control (LOAC) events, Time to the first Asthma loss of control
Acute exacerbation of severe asthma - induced hospitalization or Emergency Department visit | During 32 weeks
  Acute exacerbation of severe asthma - induced hospitalization or Emergency Department visit events
Asthma Control Questionnaire-6 (ACQ-6) score | During 32 weeks
  Mean change Mean change from baseline. The proportion of trial participants with a reduction of ≥0.5 points from baseline
Asthma Quality of Life Questionnaire (AQLQ-S) score | During 32 weeks
  Mean change from baseline
weekly Asthma Symptom Diary (ASD) score | During 32 weeks
  Mean change in mean weekly from baseline
Rescue medication | During 32 weeks
  Mean change in mean weekly from baseline
Adverse Events | During 32 weeks
Pharmacokinetics | During 32 weeks
  trough concentration
Pharmacodynamics | During 32 weeks
  mean changes of Pharmacodynamic Parameter from baseline
Anti-Drug antibody | During 32 weeks
  number and percentage of subjects tested ADA positive

CONTACTS AND LOCATIONS:
Locations (45):
- China (45):
  - Wanbei Coal-Electricity Group General Hospital, Suzhou, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Gansu Provincial People's Hospital, Lanzhou, Gansu
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Liuzhou Workers' Hospital, Liuchow, Guangxi
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Affiliated Hospital of North China University of Science and Technology, Tangshan, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The Second Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - The Third Affiliated Hospital of Qiqihar Medical University, Qiqihar, Heilongjiang
  - Anyang People's Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University, Kaifeng, Henan
  - Sanmenxia Central Hospital, Sanmenxia, Henan
  - Xinxiang First People's Hospital, Xinxiang, Henan
  - Yichang Central People's Hospital, Yichang, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Yangzhou First People's Hospital, Yangzhou, Jiangsu
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Jilin Central Hospital, Jilin, Jilin
  - Tonghua Central Hospital, Tonghua, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Ningxia Hui Autonomous Region People's Hospital, Yinchuan, Ningxia
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Heze Municipal Hospital, Heze, Shandong
  - Qilu Second Hospital of Shandong University, Jinan, Shandong
  - The Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Weifang Second People's Hospital, Weifang, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Zibo Linzi District People's Hospital, Zibo, Shandong
  - Shanghai Pulmonary Hospital (Tongji University Affiliated Shanghai Pulmonary Hospital), Shanghai, Shanghai Municipality
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Chengdu Third People's Hospital, Chengdu, Sichuan
  - Chengdu Fifth People's Hospital, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Panzhihua Integrated Traditional Chinese and Western Medicine Hospital, Panzhihua, Sichuan
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes